CLINICAL TRIAL: NCT01568164
Title: Phase II Study of the BioVentrix PliCath HF™ System for the Treatment of Ischemic Cardiomyopathy
Brief Title: Safety and Efficacy Study of the BioVentrix PliCath HF System
Acronym: CONFIGURE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioVentrix (Industry)
Collaborators: Ohio State University (Other); CDI Centro Diagnostico Italiano S.p.A (Other); Advance Research Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0015
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
Keywords: Epicardial Catheter-based Restoration; Surgical/Left Ventricular Reconstruction; Ventricular Remodeling; Dor
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device Treatment (Experimental): Treatment with the investigational device.
  Interventions: Device: PliCath HF System

INTERVENTIONS:
Device: PliCath HF System — This study is a multi-center, prospective, single-armed, study designed to evaluate the safety and efficacy of the BioVentrix PliCath HF System for left ventricular volume restoration in patients with ischemic cardiomyopathy.
  Other Names: Epicardial Catheter-based Ventricular Restoration; Dor; Surgical/Left Ventricular Reconstruction

SUMMARY:
The purpose of this prospective, single-armed, multi-center clinical trial is to further establish the safety and feasibility of using the BioVentrix PliCath HF System for the treatment of left ventricular dysfunction in appropriate cohorts of humans suffering from heart failure.

DETAILED DESCRIPTION:
Congestive heart failure is the "epidemic" of cardiovascular disease (Eugene Braunwald, NEJM 1997), yet there is no cure. The American Heart Association reports the nearly five million Americans are afflicted. Approximately 1.5 million admissions in the US are due to heart failure; it is the number one cost-item for Medicare, comprising 6% of its total expenditures.

BioVentrix has developed the PliCath heart failure system, which is used to place permanent cardiac implants into the heart for the purpose of excluding scar, reconfiguring abnormal cardiac geometry that is causing dysfunction, by excluding an abnormal portion of the ventricular wall. Conceptually, the final configuration in SVR can be achieved by placing these implants.

The procedure called PliCath Epicardial Catheter-based Ventricular Restoration System (ECVR) is designed for left ventricular volume reduction in patients with heart failure in a magnitude similar to that of the predicate surgical procedure, but much less invasively. The PliCath HF System utilizes anchors that are implanted into the scarred portion of the heart, which when deployed, exclude some of the scar similar to what is excluded by cinching the purse string suture with the patch, rendering the ventricle smaller, and is employed in a surgical setting, with and without the use of cardiopulmonary bypass.

The PliCath HF System has anchors (implants) that are deployed using fluoroscopic imaging.

ELIGIBILITY:
Inclusion Criteria

* Age 18 - 80;
* Left Ventricular Ejection Fraction (LVEF) >15% and ≤ 45%;
* NYHA FC II-IV;
* Left Ventricular End Systolic Volume (LVESVI) ≥60 cc/m² but ≤ 120 cc/ m²
* Contiguous acontractile (akinetic and/or dyskinetic) scar located in the antero-septal, apical (may extend laterally) regions of the left ventricle as evidenced by a CMR or CT;
* Maintained standard medical management for at least 90 days, and at stable target (or maximum tolerated) dosages;
* Willing and competent to complete informed consent;
* Viability of myocardium in regions remote from area of intended scar exclusion as evidenced by CMR or CT;
* Agree to required follow-up visits

Exclusion Criteria

* Calcified ventricular wall in the area of intended scar exclusion as verified by echocardiography or equivalent;
* Thrombus or intra-ventricular mass in the left atrium or ventricle as verified by echocardiography or equivalent;
* Cardiac Resynchronization Therapy (CRT) device placement ≤ 60 days prior to enrollment;
* Significant diastolic dysfunction, defined as a pseudo-normal Doppler filling pattern with E/A ratio > 2;
* Thin walled, paradoxically moving septal scar that would preclude successful support of the anchor pairs as evidenced by CMR;
* Cardiac valve disease which, in the opinion of the investigator, will require surgery;
* Intolerance or unwillingness to take anti-coagulation medication;
* Functioning pacemaker leads in antero-apical RV, which, in the opinion of the investigator, would interfere with anchor placement;
* Pulmonary Arterial Pressure > 60 mm Hg via echo;
* Myocardial Infarction within 90 days prior to enrollment;
* Previous CVA or TIA which resulted, in the opinion of the investigator, in a significant residual neurological deficit;
* Aorto iliac disease that would preclude fem-fem bypass.
* Previous right neck surgery, previous pericardiotomy, previous left chest surgery;
* Co-morbid disease process with life expectancy of less than one year;
* Patients with lung, kidney and/or liver transplant;
* Chronic renal failure with a serum creatinine >2 mg/dL;
* Pregnant or planning to become pregnant during the study;
* Enrolled in any concurrent study other than observational.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-03; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Overall rate of serious adverse events. | 24 Months
  An assessment of the overall rate of serious adverse events (SAEs) at 1 year and 2 years as adjudicated by the Data Monitoring Committee (DMC).
Primary Efficacy Endpoint - Reduction in LV Volume | 24 Months
  An assessment of measurable decrease in LV volume by either an echo or a CMR at 6 months, 1 year and 2 years.

SECONDARY OUTCOMES:
Secondary Safety Endpoint: Assessment of overall rate of serious adverse device effects. | 24 Months post operatively
  The secondary safety endpoint will be an assessment of the overall rate of serious adverse device effects (SADEs) through 2 years as adjudicated by the DMC.
Secondary Efficacy Endpoint: • Change in Left Ventricular Ejection Fraction | 24 Months
  Change in Left Ventricular Ejection Fraction (LVEF)as measured by ECHO or MRI.
Secondary Efficacy Endpoint: Hospital readmission for HF | 24 Months
  Hospital readmission for HF including surgical intervention such as Ventricular Assist Device, Cardiac Resynchronization Therapy, Intra-Aortic Balloon Pump, or transplant;
Secondary Efficacy Endpoint: Clinical utility | 24 Months
  Change in NYHA Class, Change in a standardized 6-minute corridor walk test; Change in Quality of Life (QOL) by Minnesota Living with Heart Failure (MLHF) Questionnaire.
Secondary Efficacy Endpoint: NT-proBNP | 24 Months
  Change in NT-proBNP levels

CONTACTS AND LOCATIONS:
Overall Officials: Lon Annest, MD, Study Director — Chief Medical Officer, BioVentrix
Locations (19):
- Medical University Innsbruck, Innsbruck, Austria
- NA Holmoce Hospital, Prague, Czechia
- France (2):
  - Bordeaux University Hospital Cardiology, Bordeaux
  - Hospital Pitie Sal Petirere Institute of Cardiology, Paris
- Onassis Cardiac Surgery Center, Athens, Greece
- Italy (6):
  - Spedali Civili di Cardiochirurgia, Brescia
  - IRCCS Istituto Policlinico San Donato, Milan
  - Ospedale San Raffaele, Milan
  - Padova University Hospital, Padua
  - Azienda Ospedaliera S.Camillo-Forlanini, Rome
  - Ospedale Le Molinetto, Torino
- Pauls Stradins Clinical University, Riga, Latvia
- Vilnius Hospital Santariskiu Klinikus, Vilnius, Lithuania
- Poland (2):
  - Polish American Hospital, Katowice
  - Jagiellonian University, Krakow
- CHVNGaia / Espinho Hospital, Porto, Portugal
- Hospital Clinic and University of Barcelona, Barcelona, Spain
- United Kingdom (2):
  - Kings College Hospital, London
  - The Royal Brompton Hospital, London

REFERENCES:
- [Result] Wechsler AS, Sadowski J, Kapelak B, Bartus K, Kalinauskas G, Rucinskas K, Samalavicius R, Annest L. Durability of epicardial ventricular restoration without ventriculotomy. Eur J Cardiothorac Surg. 2013 Sep;44(3):e189-92; discussion e192. doi: 10.1093/ejcts/ezt292. Epub 2013 Jun 5. PMID 23739293
- See also: Sponsor website — http://www.bioventrix.com/